CLINICAL TRIAL: NCT05832021
Title: Comparison of Patients With Distal Radius Fracture Who Underwent Surgery With WALANT Technique or Peripheral Nerve Block Anesthesia Methods in Terms of Patient Satisfaction and Functional Results in the Postoperative Period
Brief Title: Comparison of Clinical Outcomes of Distal Radius Fractures Treated Surgically With WALANT and Peripheral Nerve Block
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Huseyin Bilgehan Cevik, MD, Assoc Prof, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: 109/21
Record Dates: First submitted 2022-11-15; First posted 2023-04-27 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Distal Radius Fracture
Keywords: WALANT; Distal Radius Fracture; Peripheral nerve block
MeSH Terms: conditions — Wrist Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WALANT: Patients with distal radius fracture who underwent surgical treatment under WALANT.
  Interventions: Procedure: Open reduction and internal fixation (under WALANT)
- Peripheral nerve block: Patients with distal radius fracture who underwent surgical treatment under peripheral nerve block.
  Interventions: Procedure: Open reduction and internal fixation (under peripheral nerve block)

INTERVENTIONS:
Procedure: Open reduction and internal fixation (under WALANT) — Open reduction and internal fixation with volar Henry approach under WALANT.
  Groups: WALANT
Procedure: Open reduction and internal fixation (under peripheral nerve block) — Open reduction and internal fixation with volar Henry approach under peripheral nerve block.
  Groups: Peripheral nerve block

SUMMARY:
WALANT anesthesia technique has been frequently preferred in hand and upper extremity surgery in recent years. WALANT technique; It stands out with its advantages such as lack of pre-operative anesthesia preparation process, reduction in test and examination requests, reduction in unnecessary hospitalizations and high patient satisfaction. There are studies with a high level of evidence showing that the WALANT technique has such advantages in soft tissue and smallmedium bone fracture surgery. In large bone fractures (radius, etc.), surgical treatment is performed with the WALANT technique and positive results have been reported. Although there is a study comparing WALANT and general anesthesia in the surgical treatment of distal radius fractures, there is no study comparing the peripheral nerve block technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Patients who had acute distal radius fracture which underwent surgery

Exclusion Criteria:

* Patients with open fractures
* Additional injuries in the same extremity, peripheral vascular disease, and local anesthetic allergy at the time of first admission
* Patients who are switched to general anesthesia after both techniques
* Patients who underwent a second surgery on the same extremity due to any complication
* Patients who had lacked follow-up examination information

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 patients are planned to be included in the study.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Changes in the patient's pain | Baseline, immediately after the surgery, 2 weeks after surgery, 6 weeks after surgery, 12 weeks after surgery, 24 weeks after surgery
  Visual Analogue Scale (VAS) scale (1 to 10 score. 10 means worst pain possible, 1 is almost no pain) to measure pain level
Changes in the patient's anxiety | Baseline, immediately after the surgery, 2 weeks after surgery, 6 weeks after surgery, 12 weeks after surgery, 24 weeks after surgery
  State-Trait Anxiety Inventory (STAI-TX) (no anxiety: 1 point, a little anxiety: 2 points, anxious: 3 points, very anxious: 4 points) to measure anxiety

SECONDARY OUTCOMES:
Number of complications after surgery | Collected at end of follow up (24 months)
  Description of complications regarding surgery or anesthetical technique
Evolution in postoperative wrist mobility | Baseline, 2 weeks after surgery, 6 weeks after surgery, 12 weeks after surgery, 24 weeks after surgery
  Flexion, extension, radial and ulnar deviation, pronation and supination using a goniometer (degree)
Number of patients who need conversion to general anaesthesia due to lack of effectiveness of anaesthetic technique | During surgery (intraoperative)
  Yes or no answer to the question "did the patient need reconversion to general anaesthesia?"
Description of reason why the patient needed adding some extra anaesthesia if necessary due to lack of effectiveness of the main anaesthetic technique | During surgery (intraoperative)
  Open ended question describing the reason of anaesthesia insufficiency (for instance: pain, anxiety, discomfort, etc)
Type of anaesthetic technique added to solve the lack of effectiveness of the main anaesthesia | During surgery (intraoperative)
  Open ended question describing the technique used in order to resolve lack of anaesthesia if needed (sedation, extra doses of local anaesthetic, anatomic location of local anaesthetic, doses of local anaesthetic, etc)

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Yildirim Beyazit Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No